CLINICAL TRIAL: NCT06065982
Title: Prospective Observational Cohort Study on the Outcomes of Percutaneous Inserted PD Catheters
Brief Title: Percutaneous Peritoneal Dialysis Catheter Insertion (PREDICT)
Acronym: PREDICT
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: UMC Utrecht (Other); Leiden University Medical Center (Other); Bravis Hospital (Other); Erasme University Hospital (Other); University Hospital, Antwerp (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); az Glorieux (Unknown); Imelda Hospital, Bonheiden (Other); Centre Hospitalier Régional de la Citadelle (Other); Rijnstate Hospital (Other); Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other); HagaZiekenhuis (Other); Bernhoven Hospital (Other); Isala (Other); Deventer Ziekenhuis (Other); Medisch Centrum Leeuwarden (Unknown); OLVG (Network); Centro Hospitalar Universitario do Algarve (Other); University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: UZB-NEF-2023-PREDICT
Record Dates: First submitted 2023-04-28; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-03

CONDITIONS: End-stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — Health-related quality of life will be measured using the 12-item Short Form (SF-12) and EQ5D-5L questionnaires. The SF-12 is summarized into two component scores, the Physical Component Score (PCS) and Mental Composite Score (MCS).

SUMMARY:
Peritoneal dialysis (PD) is the most frequent modality of home dialysis for patients with kidney failure.

Most PD catheters are placed using a laparoscopic technique. This approach requires the availability of a qualified surgeon, time in the operating theater and general anaesthesia for the patient. Thus, the laparoscopic technique is less suitable for patients with severe heart failure or multimorbidity where general anaesthesia is not possible.

PD catheters can also be inserted using a percutaneous strategy using a modified Seldinger technique. This strategy can be performed bedside under local anaesthesia, by the nephrologist, radiologist, a surgeon, physician assistant or qualified nurse.

The availability of the percutaneous implantation strategy of a PD catheter in a nephrology center may accomodate more patients to receive a PD catheter insertion, including those who have a contraindication to general anaesthesia or need urgent PD.

The PREDICT project aims to increase knowledge and competencies on percutaneous PD catheter insertions by training centers for this technique. By establisching a prospective registry, the outcomes of percutaneously inserted PD catheters, both in experienced and newly trained centers, will be assessed.

DETAILED DESCRIPTION:
The population of the PREDICT study are adult patients requiring a peritoneal dialysis catheter insertion. Decision for percutaneous strategy of catheter insertion (versus surgical catheter insertion) is made by the treating physician.

The inclusion criteria for the prospective PREDICT registry are age > 18 years and percutaneous PD catheter insertion between 1 March 2023 and 1 March 1 2026 in participating centers.

Patients can be included 4 weeks before until 12 weeks after PD catheter insertion. The exclusion criteria are the inability to give informed consent and a life expectancy of less than 3 months.

Demographic and clinical data will be collected for all included patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Percutaneous PD catheter insertion between March 1st 2023 and March 1st 2026 Patients can be included 4 weeks before until 12 weeks after PD catheter insertion

Exclusion Criteria:

* Inability to provide informed consent
* Life expectancy < 3 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients requiring a peritoneal dialysis catheter insertion
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2027-06-23 (Estimated)

PRIMARY OUTCOMES:
Implementation of percutaneus PD catheter insertion technique in dialysis centers | through study completion, 3 years
  The first co-primary outcome measure assesses the implementation of the percutaneous PD catheter insertion technique in additional dialysis centers.
Outcomes of percutaneous inserted PD catheters in participating centers | Over 12 months after percutaneous insertion
  The second co-primary outcome measure assesses the outcomes of percutaneous inserted PD catheters in participating centers: functionality of PD catheters, defined as catheters usable for PD, over 12 months after percutaneous insertion, and taking into account competing events.

SECONDARY OUTCOMES:
The presence of functioning PD catheter | Over 3 and 6 months after percutaneous PD catheter insertion
  This secondary outcome measure assesses the presence of functioning PD catheter, defined as catheters usable for PD, over 3 and 6 months after percutaneous PD catheter insertion, censored for competing events.
Insertion-related complications | Perforation during or within 48 hours after catheter insertion, bleeding within 7 days of insertion, and PD-related infections within 30 days of insertion
  This secondary outcome measure assesses insertion-related complications, defined as perforation during or within 48 hours after catheter insertion, bleeding within 7 days of insertion and necessitating blood transfusion and/or invasive intervention to control bleeding, and PD-related infections (i.e. exit-site infection, tunnel infection, peritonitis) within 30 days of insertion.
Mechanical complications | through study completion of the subject, at 1 year or censored for death or kidney replacement modality switch
  This secondary outcome measure assesses mechanical complications over 3, 6, and 12 months after percutaneous PD catheter insertion. Relevant mechanical complications are defined as flow restrictions, pericatheter leakage, and abdominal pain resulting in an adverse event that is either a lack of PD start, a delay in PD start, an interruption of PD, a permanent termination of PD, emergency room visits, hospital admissions, or need for invasive procedures related to the mechanical catheter complication.
The rate of PD utilization | through study completion of the subject, at 1 year or censored for death or kidney replacement modality switch
  This secondary outcome measure assesses the rate of PD utilization, defined as 4 consecutive weeks of PD, after percutaneous PD catheter insertion, censored for competing events.
Health-related quality of life as assessed by the SF-12 questionnaire | At baseline and at 12 months after percutaneous PD catheter insertion
  This secondary outcome is assesses health-related quality of life using patient-reported outcome measures (PROMs) at baseline and at 12 months after percutaneous PD catheter insertion, using the validated SF-12 questionnaire.
Self-assessed health-related quality of life using the EQ5D questionnaire. | At baseline and at 12 months after percutaneous PD catheter insertion
  This secondary outcome is assesses health-related quality of life in terms of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using the validated EQ5D questionnaire.
Health care professionals' perspective on the implementation process | At baseline and yearly
  This secondary outcome assesses the health care professionals' perspective on the implementation process using the structured Measurement Instrument for Determinants of Innovations. This assessment allows to identify barriers and facilitators of implementation at the level of the percutaneous catheter insertion procedure, at the level of the operator and at the level of the organisation, i.e. the hospital.
Evolution in HD/PD ratio in participating centers throughout the study period | Through study completion, 3 years
  This secondary outcome assesses the evolution in HD/PD ratio in participating centers throughout the study period.
Costs of the procedure | immediately after the intervention
  The secondary outcome assesses the costs of the procedure.

CONTACTS AND LOCATIONS:
Locations (2):
- Universitair Ziekenhuis Brussel, Brussels, Belgium
- UMC Utrecht, Utrecht, Netherlands